CLINICAL TRIAL: NCT03228355
Title: The Effects of Levcromakalim on Cerebral Hemodynamic in Migraine Patients
Brief Title: Headache Inducing Effect of Cromakalim in Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Mohammad Al-Mahdi Al-Karagholi, MD, PhD student, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Levcromakalim
Record Dates: First submitted 2017-07-08; First posted 2017-07-24 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Headache, Migraine
Keywords: Levcromakalim
MeSH Terms: conditions — Migraine Disorders | interventions — Cromakalim; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levcromakalim (Active Comparator)
  Interventions: Drug: Levcromakalim
- Saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Levcromakalim — To investigate the role of Levcromakalim on cerebral hemodynamic in migraine patients
  Arms: Levcromakalim
Drug: Saline — To investigate the role of levcromakalim compared with saline cerebral hemodynamic in migraine patients.
  Arms: Saline

SUMMARY:
To investigate the role of KATP channels on the cerebral hemodynamic in migraine patients.

ELIGIBILITY:
Inclusion Criteria:

* Migraine patients of both sexes.
* 18-60 years.
* 50-90 kg.
* Women of childbearing potential must use adequate contraception.

Exclusion Criteria:

* Headache less than 48 hours before the tests start
* Daily consumption of drugs of any kind other than oral contraceptives
* Pregnant or nursing women.
* Cardiovascular disease of any kind, including cerebrovascular diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Cerebral hemodynamic | Before (-10 min) and after infusion (+2 hours) of levcromakalim compared with before and after infusion of saline
  Change on Media cerebri arterie.
Headache | Before (-10 min) and after infusion (+12 hours) of levcromakalim compared with before and after infusion of saline
  Occurrence of headache.
Migraine attack | Before (-10 min) and after infusion (+12 hours) of levcromakalim compared with before and after infusion of saline
  Occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, Professor, Study Director — DHC
Locations (1):
- Danish headache center, Copenhagen, Glostrup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Karagholi MA, Hansen JM, Guo S, Olesen J, Ashina M. Opening of ATP-sensitive potassium channels causes migraine attacks: a new target for the treatment of migraine. Brain. 2019 Sep 1;142(9):2644-2654. doi: 10.1093/brain/awz199. PMID 31292608